CLINICAL TRIAL: NCT06201065
Title: Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Plus Lenvatinib and Toripalimab Versus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Plus Lenvatinib for Advanced Hepatocellular Carcinoma: a Phase 3, Randomized Controlled and Double-blind Trial
Brief Title: FOLFOX-HAIC Plus Lenvatinib and Toripalimab vs. FOLFOX-HAIC Plus Lenvatinib for Advanced Hepatocellular Carcinoma: a Randomized Controlled and Double-blind Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SA23
Record Dates: First submitted 2023-12-25; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Lenvatinib; Oxaliplatin, Fluorouracil and Leucovorin; Hepatic arterial infusion chemotherapy; Toripalimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; toripalimab; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Hepatic arterial infusion chemotherapy plus lenvatinib and toripalimab
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Toripalimab; Drug: oxaliplatin , fluorouracil, and leucovorin
- Control arm (Active Comparator): Hepatic arterial infusion chemotherapy plus lenvatinib
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: oxaliplatin , fluorouracil, and leucovorin

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing
Drug: Toripalimab — 240 mg iv.drip Q3W
  Arms: Experimental arm
Drug: oxaliplatin , fluorouracil, and leucovorin — FOLFOX-HAIC

SUMMARY:
Our previous study showed that hepatic arterial infusion chemotherapy plus lenvatinib and toripalimab improved the survival of advanced hepatocellular carcinoma. However, Leep 002 study showded that lenvatinib plus PD-1 antibody is not superior to lenvatinib alone for advanced hepatocellular carcinoma. Thus, wo conduct this study to compare hepatic arterial infusion chemotherapy plus lenvatinib and toripalimab with hepatic arterial infusion chemotherapy plus lenvatinib for advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* This study did not limit HBV DNA load. High HBV-DNA load was aollowed, but hepatitis-B patient must receive concurrent antiviral therapy.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-07-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 18 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 18 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 18 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China